CLINICAL TRIAL: NCT06638255
Title: Effects of High Positive End-expiratory Pressure Over Abdominal Venous Congestion, Visceral Edema, and Organ Dysfunction, in Mechanically Ventilated ARDS Patients: a Randomized Cross-over Study
Brief Title: Mechanical Ventilation-induced Acute Kidney Injury [AKI]
Acronym: AKI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Martín Hernán Benites Albanese, Principal Invsetigator, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 230607001
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: ARDS; Acute Kidney Injury
Keywords: ARDS; Acute Kidney Injury; Mechanical ventilation; venous congestion
MeSH Terms: conditions — Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Intervention Model Description: To test the hypothesis, a crossover clinical-experimental protocol has been designed. Clinical and physiological data will be collected from patients with ARDS undergoing protective mechanical ventilation. Patients will be randomly allocated to two clinical protocols validated for setting PEEP levels: ARDSNet (low PEEP) and LOV (high PEEP), each for a duration of 12 hours. Clinical and physiological data, advanced ultrasound assessments, organ dysfunction markers, and a complete respiratory and hemodynamic assessment will be collected. Both PEEP strategies (Low vs High PEEP) will be applied to each patient included in the study. The PEEP setting will be selected through a computerized randomization system at the beginning of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: First Low PEEP for 12 hours, then High PEEP for 12 hours (Experimental): Arm Information
  Experimental Arm Title:
  Sequential PEEP Protocol - Low and High PEEP Strategies
  Arm Description:
  Participants in this clinical trial will be randomized into one of two pre-specified sequences to receive both high and low PEEP ventilation strategies over two sequential 12-hour periods.
  Intervention for Arm 1: Participants will receive the Low PEEP protocol for the first 12-hour period, followed by the High PEEP protocol for the next 12-hour period.
  Intervention for Arm 2 (Sequence B): Patients will receive High PEEP for the first 12 hours, then Low PEEP for the next 12 hours.
  Interventions: Other: Sequence A involves administering Low PEEP for 12 hours, followed by High PEEP for 12 hours.
- Sequence B: First High PEEP for 12 hours, then low PEEP for 12 hours (Experimental): Sequence B: First High PEEP for 12 hours, then low PEEP for 12 hours
  Interventions: Other: Sequence B involves setting High PEEP for 12 hours, followed by Low PEEP for 12 hours.

INTERVENTIONS:
Other: Sequence A involves administering Low PEEP for 12 hours, followed by High PEEP for 12 hours. — Patients will first receive the Low PEEP protocol for 12 hours, followed by the High PEEP protocol for 12 hours. This sequence is randomized and part of a crossover trial design to assess the effects of both PEEP strategies.
  Description: Patients will first receive the High or LOW PEEP protocol for 12 hours, followed by the Low or HIGH PEEP protocol for 12 hours. This sequence is randomized and part of a crossover trial design to assess the effects of both PEEP strategies.
  Other Names: Secuence A: Low PEEP vs High PEEP; Secuence B: High PEEP vs Low PEEP
  Arms: Sequence A: First Low PEEP for 12 hours, then High PEEP for 12 hours
Other: Sequence B involves setting High PEEP for 12 hours, followed by Low PEEP for 12 hours. — Sequence B involves setting High PEEP for 12 hours, followed by Low PEEP for 12 hours.
  Other Names: Only PEEP setting
  Arms: Sequence B: First High PEEP for 12 hours, then low PEEP for 12 hours

SUMMARY:
Positive end-expiratory pressure (PEEP) is a fundamental tool in the management of patients with acute respiratory distress syndrome (ARDS). However, there is currently no common criterion for deciding which level of PEEP to use. In simple terms, there are two primary strategies for setting PEEP: low PEEP and high PEEP scales. Several clinical protocols have compared them, yet no significant differences in relevant clinical outcomes have been observed. The utilization of high levels of PEEP can provide multiple benefits to the respiratory system, such as improved compliance, reduced alveolar collapse, homogenization of lung parenchyma, and notably enhanced oxygenation. Preclinical studies have shown substantial reduction in ventilator-induced lung injury when high PEEP levels were compared to low PEEP levels. Given all these relevant physiological advantages of high PEEP, the question arises: why haven´t they translated into a survival benefit in randomized controlled trials? The most rational explanation is that high PEEP simultaneously induces significant adverse effects which may counteract the potential benefits.

Some adverse effects are well known, such as the risk of overdistension and hemodynamic impairment; however, these effects are easily detected at the bedside. Negative randomized trials comparing high and low PEEP have shown no evidence of a relevant role in outcomes. In this study, abdominal venous congestion will be explored as a new potential adverse effect of high PEEP, which has not yet been studied and may play a role in counteracting the benefits of high PEEP strategies. To address this question, a randomized crossover clinical study is proposed in patients with ARDS, utilizing two previously validated and globally accepted scales of PEEP. In the following sections, the concept of ventilator-induced lung injury (VILI) will first be introduced, followed by a discussion on the beneficial effects of high PEEP on lung function and VILI prevention, in contrast to the risks of overdistension and worsening of VILI. Second, the hemodynamic effects of higher PEEP levels will be analyzed. Third, the available evidence regarding the effects of PEEP on intra-abdominal blood flow will be reviewed, and its potential relationship with the concept of abdominal venous congestion, which is well-studied in chronic heart failure, will be discussed. Finally, the role of Doppler ultrasound and elastography in studying bedside abdominal venous congestion will be addressed.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS), ventilation-induced lung injury (VILI), and protective mechanical ventilation (MV) are key aspects of respiratory failure management. ARDS is an inflammatory pulmonary edema caused by alveolar and endothelial injury, characterized by a breakdown in the alveolar-capillary barrier that results in the collapse of alveolar spaces. Clinically, ARDS manifests as acute hypoxemia, bilateral X-ray infiltrates, and decreased lung compliance. A global epidemiological study identified a 10.4% prevalence of ARDS among ICU admissions, with ICU and hospital mortality rates of 35.3% and 40.0%, respectively. ARDS survivors often experience long-term morbidity affecting the cardiovascular system, nerves, muscles, and the central nervous system. During the SARS-CoV-2 pandemic, ARDS statistics surged, placing an unprecedented burden on healthcare systems worldwide.

Mechanical ventilation serves as the primary supportive therapy for ARDS but can also exacerbate lung damage, a phenomenon referred to as VILI. VILI is primarily caused by alveolar overdistension (volutrauma) due to high tidal volumes and repeated opening and closing of unstable alveoli (atelectrauma) associated with insufficient positive end-expiratory pressure (PEEP). The late 1990s saw the first clinical trials definitively showing that lower tidal volumes improved survival rates in ARDS patients, highlighting the importance of VILI in determining ARDS outcomes. VILI also triggers a biological response characterized by lung and systemic inflammation, as well as damage to distant organs (biotrauma), which explains the role of protective ventilatory strategies in preventing organ failure and mortality.

In ARDS, a significant portion of lung units becomes unstable, collapses, and is excluded from ventilation. The collapse reduces the aerated lung size, resembling what is referred to as the "baby lung." Consequently, only this small "baby lung" receives the tidal volume, making it prone to overstretching and excessive strain. Moreover, lung infiltrates are unevenly distributed, concentrating exaggerated tensions in the healthy alveoli surrounding collapsed regions. To prevent VILI, two main ventilatory strategies have been employed: reducing tidal volume to mitigate volutrauma and optimizing PEEP to decrease atelectrauma, strain, and the uneven distribution of forces. While the protective role of low tidal volume is well-established, the role of PEEP remains a subject of ongoing debate.

The Role of PEEP in Protective Mechanical Ventilation

PEEP is defined as the maintenance of positive pressure at the airway opening at the end of expiration. Since the initial description of ARDS in 1967, PEEP has been observed to improve hypoxemia in ARDS patients by preventing alveolar collapse and recruiting collapsed lung regions, thus reducing intrapulmonary shunt. Another significant effect of PEEP is the reduction of the primary mechanisms responsible for VILI: 1) increasing the size of the "baby lung" through lung recruitment, reducing lung strain and stress; 2) keeping unstable alveoli open at end-expiration, thereby reducing opening and closing; and 3) promoting more uniform ventilation to decrease lung inhomogeneities and reduce injury at the interfaces between aerated and collapsed lung tissue.

These effects are more prominent in easily recruited lungs, while the risk of alveolar overdistension and VILI increases in less recruited lungs. Over the past 50 years, various strategies for determining appropriate PEEP levels have evolved, ranging from zero end-expiratory pressure (ZEEP) to implementing super PEEP strategies. One of the most well-known approaches is the ARDSNet PEEP/FiO2 table introduced by the National Institutes of Health ARDS Network in 1995. Although widely used, this method focused primarily on managing hypoxemia rather than preventing VILI. Subsequent trials, such as the ALVEOLI trial and the LOV trial, increased PEEP levels, but none demonstrated a mortality benefit for higher PEEP strategies.

The three largest trials comparing high versus low PEEP strategies (ALVEOLI, LOV, and EXPRESS) revealed no significant differences in mortality between the groups. A likely explanation is that higher PEEP benefits patients with substantial lung recruitability but may harm those with lower recruitability, resulting in a neutral overall effect. While higher PEEP consistently improved oxygenation across trials, improvements in respiratory compliance were less consistent. Additionally, smaller clinical studies have linked high PEEP with increased vasopressor requirements and greater fluid retention. These findings underscore the complexity of PEEP's effects on both lung mechanics and systemic physiology.

Cardiocirculatory Effects of PEEP

The hemodynamic effects of PEEP are complex and manifest in various ways in individual patients. These effects can be categorized into three primary aspects: 1) A decrease in right ventricle preload: PEEP increases pressure in the right atrium, impairing venous return. As PEEP levels gradually increase, the diameter of the inferior vena cava enlarges during both inspiration and expiration, reflecting an increase in transmural pressure and a reduction in venous return. 2) An increase in pulmonary vascular resistance: PEEP also elevates right ventricle (RV) afterload, opposing RV ejection during systole, potentially increasing RV end-diastolic volume and affecting left ventricle (LV) function downstream. These effects are influenced by factors such as lung recruitment, hyperinflation, and hypoxic vasoconstriction. 3) A decrease in left ventricle output and afterload: The primary effect of PEEP on the LV is mediated by a reduction in venous return, leading to decreased LV preload and cardiac output shortly after PEEP elevation. In patients with LV dysfunction, this reduction in afterload can enhance cardiac output and reduce myocardial oxygen demand.

In patients with acute lung injury, an increase in PEEP often results in decreased venous return and cardiac output, leading to a drop in mean arterial pressure. Intravenous fluids and/or vasoconstrictors are generally required to restore cardiac output. However, the ultimate impact of these interventions on abdominal venous congestion and tissue perfusion remains inadequately defined.

Despite the long-established awareness of PEEP's negative cardiovascular effects, its influence on intra-abdominal organs has received relatively little attention. One reason for this knowledge gap could be the challenges associated with bedside assessment of abdominal vascular flow. Over recent years, this gap has been bridged by the increased use and accessibility of Doppler ultrasonography in ICU settings. Experimental data indicate that PEEP induces redistribution of blood flow to the brain, heart, adrenals, and intestines while diminishing blood flow to the liver, pancreas, and stomach. Total renal blood flow appears to be relatively unaffected, but the redistribution of intrarenal blood flow may result in kidney dysfunction. The next sections will review the effects of PEEP on hepatic, renal, and intestinal blood flow, focusing on these three organs due to their significant role in organ dysfunction in ARDS patients.

Hepatic Blood Flow: Fujita et al. demonstrated that increasing PEEP from 5 to 10 cmH2O proportionally decreased hepatic blood flow and cardiac output without changes in mean arterial pressure. Hepatic oxygen supply and venous hemoglobin saturation were also reduced. In addition, hepatic and portal venous pressures increased with elevated PEEP, and hepatic dimensions expanded by 16-19% after applying a PEEP of 10 cmH2O. In an ARDS porcine model, Kredel et al. compared groups with 5 cmH2O PEEP and higher PEEP following a recruitment maneuver. Plasma transaminases, LDH, and bilirubin were elevated in the higher PEEP group. Brienza et al. found a strong association between mechanical ventilation with PEEP and liver dysfunction (OR 4.25; p=0.006) in critically ill patients. Recently, Huette et al. reported a progressive increase in portal pulsatility index from 9% to 45% when PEEP increased from 0 to 15 cmH2O in cardiac surgery patients, indicating venous congestion.

Renal Blood Flow: The development of acute kidney injury (AKI) is a major contributor to ICU morbidity and poor long-term outcomes. PEEP has been associated with reduced renal perfusion and glomerular filtration, as well as elevated levels of antidiuretic hormone, plasma renin, and aldosterone. These changes coincide with decreased natriuresis and water retention, which can contribute to venous congestion. A comprehensive retrospective cohort study by Geri et al. linked mechanical ventilation (MV) to renal function deterioration, with PEEP playing a significant role in this association due to renal venous congestion. Dres et al. demonstrated that high PEEP correlated with higher AKI incidence and an increased need for renal replacement therapy in COVID-19 ARDS patients. In a study by Fogagnolo et al., a linear correlation was found between PEEP levels and the renal resistive index (R²=0.31; p=0.03), with 71% of patients showing non-continuous renal venous flow under high PEEP.

Intestinal Blood Flow: Lehtipalo et al. evaluated intestinal perfusion in a porcine model using invasive Doppler measurements, finding that hepatosplanchnic blood flow progressively declined as PEEP increased from ZEEP to 12 cmH2O. This was associated with a parallel increase in oxygen extraction. The effects of this maneuver were more pronounced when abdominal perfusion pressure dropped below 50 mmHg. Additionally, mechanical ventilation with positive pressure impeded lymphatic drainage from the interstitium, leading to interstitial fluid retention. In an endotoxemic porcine model, Lattuada et al. compared three groups (spontaneous ventilation, PEEP 5 cmH2O, and PEEP 15 cmH2O) and observed that increasing PEEP proportionally decreased lymphatic flow from the abdomen and increased liver and intestinal edema and inflammation. These effects were attributed to increased systemic capillary leakage and impeded abdominal lymph drainage. Experimental data suggest that PEEP-induced venous congestion in abdominal organs, resulting from reduced pressure gradients between the arterial and venous systems, leads to increased oxygen extraction, organ dysfunction, and local inflammation.

The most extensively studied pathological model of abdominal congestion is secondary to chronic global heart failure, which leads to reduced cardiac output, increased filling pressures, and fluid overload. In these patients, visceral edema can progress to severe complications such as cirrhosis, terminal renal failure, and intestinal dysfunction, with increased permeability to endotoxins and bacteria. This condition is exacerbated by a systemic inflammatory state, worsening the patient's prognosis. PEEP can induce a similar pathophysiological state through elevated right heart filling pressures, even in the absence of right ventricular dysfunction or hypervolemia. In ARDS patients, factors such as decreased oncotic pressure, increased vascular permeability due to inflammation, and elevated hydrostatic pressure (fluids and transfusions) contribute to the negative impact of venous congestion caused by PEEP. Fluid accumulation in encapsulated organs such as the liver and kidneys is poorly tolerated due to limited expansion, intensifying perfusion disturbances.

In terms of specific organ perfusion, venous congestion increases post-capillary pressure. If PEEP reduces cardiac output, precapillary pressure may also decrease, disrupting the balance between these factors and potentially leading to organ dysfunction. Doppler ultrasound (US) serves as an effective, non-invasive tool for evaluating arterial and venous abdominal vasculature, providing clinicians with valuable data on organ-specific blood flow. In recent years, US has gained prominence in assessing abdominal venous systems. The VExUS (venous excess ultrasound) score, combining multiple venous Doppler signals (inferior vena cava, hepatic vein, portal vein, and renal vein), has been validated in cardiac surgery patients and correlated with right atrial pressure (R²=0.68). In addition, VExUS has been positively associated with diuretic response and AKI development in acute coronary syndrome patients, with ongoing studies evaluating its role in post-sepsis venous congestion.

Ultrasound elastography measures tissue stiffness or elasticity and is useful in evaluating liver and kidney diseases. Kashani et al. demonstrated that ultrasound surface wave elastography correlates with transcatheter kidney intracapsular pressure measurements. This technology has multiple clinical applications, especially in detecting renal fibrosis. More recently, elastography has been shown to detect renal tissue damage in cirrhotic patients earlier than routine lab tests. Liver stiffness measured by elastography has been linked to liver congestion in models of inferior vena cava clamping and is increasingly considered a useful tool for estimating right atrial pressure and predicting diuretic response.

Integrating PEEP Setting, Abdominal Venous Congestion, Edema, and Organ Dysfunction

In summary, PEEP is considered a fundamental tool in managing ARDS patients as it improves oxygenation and, under experimental conditions, decreases the likelihood of developing VILI. However, these benefits have not been reflected in significant improvements in relevant clinical outcomes, such as reduced mortality or the duration of mechanical ventilation. There is no single rule for setting PEEP, and clinicians generally use high or low levels of PEEP based on individual preferences, balancing the benefits (oxygenation, lung protection, and mechanics) with the potential adverse effects, such as alveolar overdistension and hemodynamic compromise. PEEP can potentially decrease cardiac output and induce abdominal venous congestion by limiting venous return to the thorax. In cases of chronic heart failure, abdominal venous congestion can result in severe organ failure, such as cirrhosis and terminal renal failure, promoting a systemic inflammatory state that exacerbates the harmful effects of cardiac failure, leading to increased complications and worsening the patient's prognosis.

Given these arguments, the question arises as to whether the potential benefits of using high levels of PEEP, particularly at the pulmonary level, may be counterbalanced by adverse effects on organs outside the thorax. It is hypothesized that the use of high PEEP levels, in comparison to low levels, significantly increases abdominal venous congestion, visceral edema, and organ dysfunction in patients with moderate to severe ARDS. To explore this hypothesis, a randomized crossover clinical study has been designed to evaluate the impact of PEEP as a generator of abdominal venous congestion, edema, and organ dysfunction over a 12-hour period. This study design will allow for each intervention to be assessed within the same subject, functioning as their own control, thereby providing greater efficiency in comparing effects. It is anticipated that this study will contribute to a better identification of patients at risk of developing abdominal complications secondary to PEEP in the near future.

Hypothesis:

The use of high levels of PEEP, compared to low levels of PEEP, significantly increases abdominal venous congestion, visceral edema, and organ dysfunction in patients with moderate to severe ARDS.

General objective:

To compare the effect of applying high and low PEEP levels on respiratory mechanics, hemodynamics, abdominal venous congestion, visceral edema, and organ dysfunction in patients with moderate to severe ARDS.

Specific Objectives:

Correlate the impact of high and low PEEP levels on cardiorespiratory physiology with the degree of abdominal venous congestion.

Experimental design: Throughout the study, a comprehensive physiological and clinical assessment will be conducted, focusing on hemodynamics, respiratory mechanics, and gas exchange parameters. Continuous recordings of lung and respiratory system mechanics (respiratory compliance, lung collapse, and overdistension, bedside potential for recruitment, EIT ventilatory distribution, volumetric capnography, and ABGs) will be made. A complete hemodynamic assessment (including echocardiogram, invasive arterial and central venous pressure, and markers of tissue perfusion such as lactate, central venous saturation, and veno-arterial CO₂ gradient) will also be performed to analyze trends and absolute values. These assessments will provide insights into the impact of different PEEP strategies on patient cardiorespiratory physiology and their integration with the degree of venous congestion.

Measure the effect of high and low PEEP levels on abdominal venous congestion and visceral edema.

Experimental design: Surface Doppler ultrasound will be utilized to comprehensively analyze blood flow in the venous and arterial abdominal circulation. The primary focus will be on venous circulation, employing the VExUS protocol. Regular assessments of this parameter will be conducted every 4 hours, and at the end of each 12-hour period, a thorough ultrasonographic analysis of both arterial and venous systems will be performed, along with assessments for signs of visceral edema. Data will be collected for subsequent offline waveform pattern analysis, enabling the identification of alterations in venous flow velocity, direction, and resistance to flow. Sequential evaluations of transient elastography will also be employed to determine liver and kidney tissue changes associated with edema and congestion.

Determine the effect of abdominal venous congestion on renal, hepatic, and intestinal dysfunction.

Experimental design: Plasma levels of specific markers associated with renal (N-Gal, Cyst-C, creatinine, blood urea nitrogen, ADH, renin, aldosterone), liver (bilirubin, AST, ALT, alkaline phosphatases, and gamma-glutamyl transpeptidase), and intestinal dysfunction (plasma zonulin, calprotectin, and endotoxin levels) will be assessed and compared sequentially. Additionally, some renal dysfunction markers will be monitored sequentially in urine plus urinary sediment to detect early changes in tubular function. The response of the renin-angiotensin-aldosterone axis to hemodynamic changes will also be examined.

Scientific or Technological Novelty of the Proposal:

Traditionally, the impact of PEEP on the cardiovascular system has focused on cardiac function (both right and left), and it is considered well-tolerated if macrohemodynamics (e.g., systemic blood flow and blood pressure) are maintained within clinically acceptable ranges. However, this approach may be considered incomplete, as the use of high PEEP levels affects the entire system, requiring adaptation to unusual pressure ranges, which results in flow redistribution and subdiaphragmatic venous congestion. This study aims to fill this knowledge gap by focusing on the effects of PEEP on venous circulation, perfusion, and abdominal organ function. The goal is to unveil physiological elements that help to explain why, despite consistently improving oxygenation and respiratory mechanics, the use of high PEEP levels has not demonstrated improvements in clinically relevant outcomes, such as mortality or length of stay. Depending on the results, PEEP regulation may be considered based not only on respiratory outcomes or cardiopulmonary interaction but also on a thoracoabdominal perspective.

From a technological standpoint, this proposal is innovative as it introduces clinical and ultrasonographic monitoring of abdominal circulation and visceral edema. The VExUS system will be employed for these purposes, which have previously been validated in the evaluation of post-cardiac surgery patients but never for the monitoring of ARDS patients. If VExUS proves useful in this evaluation, a new non-invasive hemodynamic monitoring method for ARDS patients could be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and severe ARDS, as defined by the Berlin Definition
* Connection to mechanical ventilation for less than seven days

Exclusion Criteria:

* Acute respiratory failure due to exacerbation of chronic respiratory disease or cardiogenic pulmonary edema
* Acute or chronic hepatic failure
* Chronic renal failure
* Acute renal failure (KDIGO Stage 3)
* Patients with a decision not to resuscitate
* Critically ill patients who are unable to tolerate ventilatory changes
* Patients in the prone position

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Elevation of plasma and urinary biomarkers of acute kidney injury (NGAL - KIM-1) | 12 hours
  Elevation of plasma and urinary biomarkers of acute kidney injury associated with high PEEP strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
The variables of interest will be shared to an extent reasonable.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Gattarello S, Lombardo F, Romitti F, D'Albo R, Velati M, Fratti I, Pozzi T, Nicolardi R, Fioccola A, Busana M, Collino F, Herrmann P, Camporota L, Quintel M, Moerer O, Saager L, Meissner K, Gattinoni L. Determinants of acute kidney injury during high-power mechanical ventilation: secondary analysis from experimental data. Intensive Care Med Exp. 2024 Mar 21;12(1):31. doi: 10.1186/s40635-024-00610-1. PMID 38512544
- [Background] Beurton A, Haudebourg L, Simon-Tillaux N, Demoule A, Dres M. Limiting positive end-expiratory pressure to protect renal function in SARS-CoV-2 critically ill patients. J Crit Care. 2020 Oct;59:191-193. doi: 10.1016/j.jcrc.2020.07.008. Epub 2020 Jul 10. No abstract available. PMID 32683213
- [Background] Fogagnolo A, Grasso S, Dres M, Gesualdo L, Murgolo F, Morelli E, Ottaviani I, Marangoni E, Volta CA, Spadaro S. Focus on renal blood flow in mechanically ventilated patients with SARS-CoV-2: a prospective pilot study. J Clin Monit Comput. 2022 Feb;36(1):161-167. doi: 10.1007/s10877-020-00633-5. Epub 2021 Jan 1. PMID 33385260
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Background] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162